CLINICAL TRIAL: NCT04571645
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Dociparstat Sodium in Combination With Standard Chemotherapy for the Treatment of Newly Diagnosed Acute Myeloid Leukemia
Brief Title: Dociparstat in Combination With Standard Chemotherapy for the Treatment of Acute Myeloid Leukemia
Acronym: AML
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study enrollment was terminated on 16 May 2022 due to slow recruitment.
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMX-DS-003
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Results first posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dociparstat (Experimental): Treatment with standard intensive induction, reinduction, or consolidation chemotherapy and dociparstat 4 mg/kg intravenous (IV) bolus on Day 1, administered 30 minutes after completion of the first dose of idarubicin or daunorubicin, followed by dociparstat 0.25 mg/kg/hr via continuous IV infusion 24 hours daily for 5 or 7 days.
  Interventions: Drug: Dociparstat
- Control (Placebo Comparator): Treatment with standard intensive induction, reinduction, or consolidation chemotherapy and placebo intravenous (IV) bolus on Day 1, administered 30 minutes after completion of the first dose of idarubicin or daunorubicin, followed by placebo via continuous IV infusion 24 hours daily for 5 or 7 days.
  Interventions: Other: Control

INTERVENTIONS:
Drug: Dociparstat — Dociparstat is a glycosaminoglycan derived from porcine heparin.
  Other Names: DSTAT; CX-01; 2-0,3-0 desulfated heparin; ODSH; dociparstat sodium
  Arms: Dociparstat
Other: Control — 0.9% Normal Saline
  Other Names: 0.9% Normal Saline; Normal saline; Sodium chloride 0.9%
  Arms: Control

SUMMARY:
Phase 3 study to evaluate the efficacy and safety of dociparstat sodium in adults with newly diagnosed untreated acute myeloid leukemia (AML) with adverse or intermediate genetic risk.

DETAILED DESCRIPTION:
A Phase 3, multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of dociparstat sodium in combination with standard intensive induction and consolidation chemotherapy for the treatment of newly-diagnosed acute myeloid leukemia (AML) patients.

ELIGIBILITY:
Inclusion Criteria:

A potential participant must have met all the following criteria to be eligible to participate in the study:

1. Had newly-diagnosed, previously untreated acute myeloid leukemia (AML) (according to the World Health Organization criteria) with at least 20% blasts in the peripheral blood or bone marrow.
2. Was aged ≥18 years.

   1. Adverse genetic risk (according to European LeukemiaNet [ELN] criteria), defined as nay of the following genetic abnormalities:

      * t(6;9)(p23;q34.1); DEK-NUP214
      * - t(v;11q23.3); KMT2A rearranged
      * - t(9;22)(q34.1;q11.2); BCR-ABL1
      * - inv(3)(q21.3q26.2) or t(3;3)(q21.3;q26.2); GATA2, MECOM(EVI1)
      * - -5 or del(5q); -7; -17/abn(17p)
      * - Complex karyotype, monosomal karyotype
      * - Wild-type NPM1 and FLT3-ITDhigh
      * - Mutated RUNX1, mutated ASXL1, or mutated TP53 OR
   2. Intermediate genetic risk (according to ELN criteria), defined as any of the following genetic abnormalities:

      * Mutated NPM1 and FLT3-ITDhigh
      * - Wild-type NPM1 without FLT3-ITD or with FLT3-ITDlow (without adverse-risk genetic lesions)
      * - t(9;11)(p21.3;q23.3); MLLT3-KMT2A
      * - Cytogenetic abnormalities not classified as favorable or adverse
3. Had an Eastern Cooperative Oncology Group performance status of 0 to 2.
4. Provided written informed consent to participate in the study.

Exclusion Criteria:

A potential participant who met any of the follow criteria was not eligible to participate in the study:

Leukemia exclusions:

1. Had acute promyelocytic leukemia (t(15;17)), myeloid sarcoma without bone marrow involvement, or blast transformation of chronic myelogenous leukemia.
2. Not applicable (criterion removed in Amendment 1 of the Clinical Study Protocol).
3. Not applicable (criterion removed in Amendment 1 of the Clinical Study Protocol).
4. Had clinical evidence of central nervous system leukemia.

   Prior/Concomitant Therapy:
5. Had previously received AML treatment, including Vyxeos (CPX-351, liposomal cytarabine and daunorubicin), gemtuzumab ozogamicin, or any other prohibited concomitant AML therapy previously received or anticipated to start during the study.

   Note: Prior hydroxyurea and emergency leukapheresis to control white blood cell count were allowed. All-trans retinoic acid during workup and a single dose of intrathecal cytarabine and/or methotrexate was permitted for participants who were undergoing lumbar puncture to evaluate central nervous system involvement.
6. Were receiving any form of anticoagulant therapy (e.g., unfractionated heparin, low molecular weight heparin, coumadin, factor Xa inhibitors).

   Note: Heparin flush of indwelling catheters was permitted.
7. Received treatment with any other investigational agent within 28 days or 5 half-lives, whichever was longer, prior to baseline.
8. Underwent any major surgery or radiation therapy within 28 days prior to baseline.

   Medical conditions:
9. Had immediately life threatening, severe complications of leukemia such as pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation.
10. Had active or uncontrolled bleeding at the time of randomization; a bleeding disorder, either inherited or caused by disease; a history of known arterial-venous malformation, intracranial hemorrhage, or suspected or known cerebral aneurysm; or clinically significant (in the judgement of the Investigator) gastrointestinal bleeding within 3 weeks prior to randomization.
11. Had the presence of significant active or uncontrolled infection, including human immunodeficiency virus (HIV) or hepatitis B or C.

    Note: Subjects with an infection who were receiving treatment (antibiotic, antifungal, or antiviral treatment) may have entered into the study but must have been afebrile and hemodynamically stable for ≥72 hours. Patients who had current evidence of invasive fungal infection (positive blood or tissue culture) must have had subsequent negative cultures to be eligible.
12. Had active (uncontrolled, metastatic) second malignancy. Note: A second malignancy that was in remission was permitted if there was clinical evidence of disease stability for a period of greater than 6 months off cytotoxic chemotherapy that was documented by imaging, tumor marker studies, etc. Long-term nonchemotherapy treatment (e.g., hormonal therapy) was acceptable.
13. Had psychiatric or neurological conditions that could have compromised participant safety or compliance.
14. Had a history of severe congestive heart failure or other cardiac disease that contraindicated the use of idarubicin or daunorubicin (e.g., cardiac ejection fraction <45%, as determined by echocardiography or multigated acquisition scan).

    Diagnostic assessments:
15. Had a corrected QT interval >480 msec.
16. Had severe renal impairment, as determined by calculated creatinine clearance <30 mL/min or estimated glomerular filtration rate <30 mL/min/1.73 m2.
17. Had alanine aminotransferase or aspartate aminotransferase >3x the upper limit of normal (ULN) or total bilirubin >2x the ULN.

    Other:
18. Was a woman of childbearing potential who was pregnant, breastfeeding, and/or not using a highly effective method of contraception (consistent with local regulations regarding the methods of contraception for those participating in clinical studies).
19. Had a history of allergy or hypersensitivity to heparin, pork, or any excipients in the dociparstat formulation.
20. Had any other condition, including abnormal laboratory values that, in the judgement of the Investigator, could have put the participant at increased risk or interfered with the conduct or planned analyses of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - UC Irvine Medical Center, Orange, California
  - University of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute, St. Matthews Campus, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Henry Ford Health System, Detroit, Michigan
  - Allina Health System / Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - New York Medical College, Hawthorne, New York
  - Mount Sanai School of Medicine, New York, New York
  - East Carolina University Vidant Medical Center, Greenville, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Spartanburg Medical Gibbs Cancer Center, Spartanburg, South Carolina
  - Baylor, Dallas, Texas
  - University of Utah / Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dociparstat Sodium (DSTAT): Treatment with standard intensive induction, reinduction, or consolidation chemotherapy and Dociparstat 4 mg/kg IV bolus on Day 1, administered 30 minutes after completion of the first dose of idarubicin or daunorubicin, followed by Dociparstat 0.25 mg/kg/hr via continuous IV infusion 24 hours daily for 5 or 7 days.
  Dociparstat sodium: Dociparstat is a glycosaminoglycan derived from porcine heparin.
- Control: Treatment with standard intensive induction, reinduction, or consolidation chemotherapy and Placebo IV bolus on Day 1, administered 30 minutes after completion of the first dose of idarubicin or daunorubicin, followed by Placebo via continuous IV infusion 24 hours daily for 5 or 7 days.
  Placebo: 0.9% Normal Saline
Period: Overall Study
Arm/Group | Dociparstat Sodium (DSTAT) | Control
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dociparstat Sodium (DSTAT) | Control | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Median (Full Range); unit: years] | 67 [61 to 69] | 64 [47 to 65] | 65 [47 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined for all study participants through 5 years after randomization.
  Overall survival was to be measured from the date of randomization to the date of death from any cause. Participants not known to have died at last follow-up contact were to be censored on the date they were last known to be alive.
  Due to early termination, subjects did not complete long term follow-up and efficacy (including overall survival outcome) was not analyzed.
Time Frame: Measured from randomization to date of death from any cause, up to 1 year.
Population: Due to the early termination of the study, efficacy (overall survival) was not formally analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Dociparstat Sodium (DSTAT) | Control
Number analyzed (Participants) | 5 | 4
Participants | 4 | 4

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed through study completion, up to 1 year; all adverse events were collected through 42 days after the start of the last cycle of study intervention, up to 168 days.
Description: Adverse events were collected in all subjects from the time of the first dose through 42 days after the start of the last cycle with study intervention (i.e., dociparstat or placebo administered during initial induction, reinduction, or consolidation therapy).
Arm/Group | Dociparstat Sodium (DSTAT) | Control
All-Cause Mortality (participants affected / at risk) | 1/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 3/5 | 1/4
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dociparstat Sodium (DSTAT) (N=5) | Control (N=4)
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dociparstat Sodium (DSTAT) (N=5) | Control (N=4)
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Enteritis (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Glossitis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 1
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Catheter site rash (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 2
Pyrexia (General disorders) | 0 | 2
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0
Adenovirus infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Blood albumin decreased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Brain natriuretic peptide increased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 2
Platelet count decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 1
Hallucination (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to low subject accrual, study enrollment was prematurely terminated on 16 May 2021. Therefore, formal statistical analyses were not performed, and no conclusions can be drawn about dociparstat with regards to efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 18 months of the completion of the Study at all sites, if no publication of the overall multi-center results has been made, institutions are entitled to publish their locally obtained results, provided the Sponsor is given opportunity to review and comment. Institution publications may be delayed up to an additional 60 days to allow Sponsor to seek patent protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT04571645/Prot_SAP_000.pdf